CLINICAL TRIAL: NCT04141865
Title: Effect of Xen Implantation on the Aqueous Humor Proteome
Status: Terminated | Type: Observational
Why Stopped: low enrollment
Sponsor: Price Vision Group (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-006
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Glaucoma Drainage Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Aqueous humor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Xen: Patients treated with a Xen microstent for glaucoma.
  Interventions: Device: Xen
- Aqueous shunt: Patients treated with an aqueous shunt for glaucoma.
  Interventions: Device: Aqueous shunt

INTERVENTIONS:
Device: Xen — Xen microstent implantation
  Groups: Xen
Device: Aqueous shunt — Aqueous shunt implantation
  Groups: Aqueous shunt

SUMMARY:
The purpose of this study is to determine how the aqueous humor proteome changes after implantation of a Xen microstent for treatment of glaucoma.

DETAILED DESCRIPTION:
The purpose of this study is to determine how the aqueous humor proteome changes after implantation of a Xen microstent for treatment of glaucoma using liquid chromatography mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any racial or ethnic origin, 18 years or older
* Able to provide written informed consent.
* Scheduled to undergo Xen implantation for open angle glaucoma or already has an aqueous shunt

Exclusion Criteria:

* History of conjunctivitis or any ocular infection within the past 3 weeks.
* Any active inflammation of the cornea or the anterior chamber (uveitis)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with open angle glaucoma treated with a glaucoma drainage device.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Aqueous humor proteome | Change from baseline at 6 months
  The aqueous humor proteome will be assessed with liquid chromotography/mass spectometry (quantitative LC-MS/MS).

CONTACTS AND LOCATIONS:
Overall Officials: Francis Price, Jr, MD, Principal Investigator — Price Vision Group
Locations (1):
- Price Vision Group, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
de-identified data will be available upon request